CLINICAL TRIAL: NCT01406470
Title: An Open-Label, Single-Arm, Historically Controlled, Prospective, Multicenter Phase III Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Immune Globulin Intravenous (Human) IVIG-SN™ in Subjects With Primary Immunodeficiency
Brief Title: Phase 3 Study of Immune Globulin Intravenous (Human)IVIG-SN™ in Subjects With Primary Immunodeficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIG_SN_P3; IVIG_SN_P3 (Other Grant/Funding Number: Green Cross Corporation)
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Immunologic Deficiency Syndrome
Keywords: IGIV; Primary Immune Deficiency; Immunoglobulin G
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVIG-SN™ (Experimental): Immune Globulin Intravenous (Human) 5% Liquid
  Interventions: Drug: Immune Globulin Intravenous (Human) 5% Liquid, IVIG-SN™

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human) 5% Liquid, IVIG-SN™ — IVIG-SN™ 10g/200mL, dose is 300-900 mg/kg/infusion every 21 or 28 days, intravenously. The total duration of treatment with IVIG-SN™ will be 12 months with a 3 month follow-up.
  Other Names: IGIV; Immune Globulin Intravenous (Human) 5% Liquid

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics of Immune Globulin Intravenous (Human) IVIG-SN™ in subjects with primary immunodeficiency diseases.

DETAILED DESCRIPTION:
This is an open-label, single-arm, historically controlled, prospective, multicenter phase III study to evaluate the safety, efficacy and pharmacokinetics of Immune Globulin Intravenous (Human) IVIG-SN™ in subjects with primary immunodeficiency diseases.

Subject will be infused every 21 to 28 days according to their previous IVIG treatment schedule. Subjects treated every 28 days will receive 13 study IVIG infusions. Subject treated every 21 days will receive 17 study IVIG infusions.

Duration of treatment:The total duration of treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed clinical diagnosis of a Primary Immunodeficiency Disease as defined by IUIS (International Union of Immunological Societies) and require treatment with IVIG. Documented agammaglobulinemia or hypogammaglobulinemia (preferably with documented antibody deficiency).
* Male or female, ages 2 to 70 years.
* The subject has received 300-900 mg/kg of a licensed IGIV therapy at 21 or 28 day intervals for at least 3 months prior to this study.
* At least 2 documented IgG trough levels of ≥ 5 g/L are obtained at two infusion cycles (21 or 28 days) within 12 months prior to study enrollment.
* Subject is willing to comply with all requirements of the protocol.
* Females of child-bearing potential with a negative urine pregnancy test and who agree to employ adequate birth control measures during the study.
* Subject, parent or guardian has signed the informed consent form and a child assent form if appropriate. Pediatric subjects are defined as 2-17 years of age at study entry and will require assent forms as appropriate per study documentation and regulations of the local jurisdiction.
* Authorization to access personal health information.
* Subjects currently participating in a clinical trial with another experimental IVIG may be enrolled if they have received stable IVIG therapy for at least 3 infusion cycles prior to receiving IVIG-SN™ and all inclusion and exclusion criteria are satisfied. Other IVIGs will be prohibited between the first infusion of IVIG-SN™ and Follow Up Visit 1.
* Subjects currently participating in a trial of SCIG can be enrolled if they are switched to IVIG for three infusion cycles (21 or 28 days) prior to enrollment in this study.

Exclusion Criteria:

* Subject has secondary immunodeficiency.
* Subject was newly diagnosed and has not been treated with immunoglobulin or has been diagnosed with dysgammaglobulinemia or isolated IgG subclass deficiency.
* Subject has a history of repeated reactions or hypersensitivity to IVIG or other injectable forms of IgG.
* Subject has a history of thrombotic events including deep vein thrombosis, cerebrovascular accident, pulmonary embolism or transient ischemic attacks, or myocardial infarction, as defined by at least 1 event in subject's lifetime.
* Subject has IgA deficiency and is known to have antibodies to IgA.
* Subject has received blood products other than human albumin or human immunoglobulin within 12 months prior to enrollment.
* Subject has significant protein losing enteropathy, nephrotic syndrome or lymphangiectasia.
* Subject has an acute infection as documented by culture or diagnostic imaging and/or a body temperature exceeding 38.5 °C (101.3 °F) within 7 days prior to screening
* Subject has a known history or is positive at enrollment for human immunodeficiency virus (HIV) type 1/2 by NAT or hepatitis B virus (HBsAg and NAT) or hepatitis C virus (by NAT), or hepatitis A virus (by NAT).
* Subject has levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times of the upper limit of normal for the laboratory designated for the study.
* Subject is using an implanted venous access device
* Subject has profound anemia or persistent severe neutropenia (≤ 1000 neutrophils per mm3).
* Subject has a severe chronic condition such as renal failure (creatinine concentration > 2.0 times the upper limit of normal) with proteinuria, congestive heart failure (New York Heart Association III/IV), cardiomyopathy, cardiac arrhythmia associated with thromboembolic events (e.g. atrial fibrillation), unstable or advanced ischemic heart disease, or hyperviscosity, or any other condition that the investigator believes is likely to interfere with evaluation of the study drug or with satisfactory conduct of the trial.
* Subject has a history of a malignant disease other than properly treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin within 24 months prior to enrollment.
* Subject has history of epilepsy or multiple episodes of migraine not completely controlled by medication.
* Subject is receiving the following medication:

  * Steroids (oral or parenteral daily dose of ≥ 0.15 mg/kg/day of prednisone or equivalent).
  * Other immunosuppressive drugs or chemotherapy.
* Females who are pregnant, breast feeding or planning a pregnancy during the course of the study. Women who become pregnant during the study will be withdrawn from the study.
* Subject has participated in another clinical study within 3 weeks prior to study enrollment.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of acute serious bacterial infections | one year
Overall incidence of adverse events that occur during or within 1 hour, 24 hours and 72 hours following an infusion of test product | Within 72 hours after treatment with IVIG-SN
The Pharmacokinetic (PK) Area under the curve (AUC0-t, AUC0-inf) of Immunoglobulin G (IgG). | After 5th infusion
The Pharmacokinetic (PK) Maximum concentration (Cmax) of Immunoglobulin G (IgG). | After 5th infusion

SECONDARY OUTCOMES:
The number of days missed work/school/kindergarten/day care or unable to perform normal daily activities due to infection. | one year
Days of unscheduled physician visits and hospitalizations due to infection | One year
Number of days on therapeutic antibiotics | One year
The incidence of infections other than acute serious bacterial infections | One year
Annual rate of fever episodes per patient | One year
All adverse events regardless of causality assessment by investigator | One year
The proportion and number of IGIV infusions for which the infusion rate was decreased due to adverse events | One year
The proportion of adverse events considered by the investigator to be product related | One year
To monitor viral safety (freedom from transmission of blood borne virus diseases) | One year
Descriptive analyses of PK parameters for specific antibodies (anti-Hemophilus influenza type b, anti-Streptococcus pneumonia serotypes, anti-Tetanus toxoid, anti-cytomegalovirus (CMV), anti-measles) will be performed. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Roifman, MD, Study Chair — The Hospital for Sick Children
Locations (11):
- United States (9):
  - University of Alabama Hospital, Birmingham, Alabama
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Optimed Research, LTD, Columbus, Ohio
  - Dallas Allergy Immunology, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - Children's Hospital of Richmond, Richmond, Virginia
  - Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington
- Canada (2):
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario